CLINICAL TRIAL: NCT05902130
Title: Symptoms of Acute Coronary Syndrome in Medical Regulation: a Retrospective Study
Brief Title: Symptoms of Acute Coronary Syndrome in Medical Regulation
Acronym: SCAST+
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-03Obs-CHRMT
Record Dates: First submitted 2023-05-22; First posted 2023-06-13 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; out-hospital care; medical regulation
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: symptoms of a myocardial infarction — Analysis of the differences in symptoms of a myocardial infarction between a man and a woman

SUMMARY:
The main objective was to analyze the impact of the gender of the attending physician in the differences in the management of ST+ ACS between men and women.

This study will be conducted in partnership with the interventional cardiology team of the CHR Metz-Thionville and SAMU (emergency call center) of Moselle, which has a detailed registry of coronary angiographies at the center. A retrospective observational study will be carried out over a "typical" period outside of covid at the CHR Metz Mercy (2021-2022) based on coronary angiographies performed in the context of ST+ ACS at the CHR of patients referred by the center 15.

The patient's medical record will be analyzed, going back to his call to the 15 via tape listening. The number of subjects required being calculated at 104 men and 104 women, these patients will be selected from the database of our cardiologist colleagues and we will match one man to one woman by comparing the delays of several items (1st medical contact, time of 1st ECG, medicalization or not, delay of call to the cardiologist, delay of coronary angiography...) according to the sex of the regulator. The consequences of a difference in management will be also evaluated by analyzing in-hospital mortality, mortality at 30 days of management, and functional sequelae at discharge (grades of dyspnea, disturbance of myocardial contractility, LVEF at discharge).

This study based on the differences in questioning according to the gender of the regulating physician would allow better identification of the factors that increase the delay in the management of ST+ ACS in women, and to find avenues of correction in order to limit the loss of opportunity for patients.

The patients included who are still alive will receive a notification of non-objection by mail.

ELIGIBILITY:
Inclusion Criteria:

* patient with emergency coronary angiography for ST+ ACS
* having made a call to the Emergency Center for the same reason

Exclusion Criteria:

* non-real ST+ ACS

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The cohort includes patients admitted for coronary angiography at the Mercy hospital center in 2021-2022, having had a confirmed diagnosis of ACS ST+ and who made an initial call to the Moselle SAMU.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Delay between the call to the emergency center and the first contact with a physician | End of the call to the emergency center, less than 10 min
  Delay (minutes:seconds)

SECONDARY OUTCOMES:
Delay between the call to the emergency center and the first electrocardiogram | At hospital discharge, an average of 2 hours
  Delay (hours:minutes)
Dispatch of a medical ambulance (Y/N) | End of the call to the emergency center, an average of 20 min
  Number (%)
Delay between the call to the emergency center and the first coronary angiography | At hospital discharge, an average of 2 hours
  Delay (minutes)
In-hospital mortality | 30 days after the call to emergency center
  Number (%)
Day 30 mortality | 30 days after the call to emergency center
  Number (%)
Left Ventricular Ejection Fraction | At hospital discharge, less than 30 days
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Laure ABENSUR VUILLAUME, MD, PhD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No